CLINICAL TRIAL: NCT04500067
Title: An Open-label Multicenter Randomized Trial to Evaluate the Efficacy of Bioven, Manufactured by Biopharma Plasma, LLC, in Complex Therapy of Patients With Pneumonia Induced by COVID-19 / SARS-CoV-2
Brief Title: Intravenous Immunoglobulin (IVIG, Bioven) Efficacy Assess for COVID-19 / SARS-CoV-2 Severe Pneumonia Complex Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biopharma Plasma LLC (Industry)
Collaborators: Lviv National Medical University (Other); Vinnitsa National Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-BV-BP
Record Dates: First submitted 2020-07-15; First posted 2020-08-05 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Covid19; Pneumonia
Keywords: Pneumonia; COVID-19; SARS-CoV-2; IVIG; Immunoglobulin for Intravenous Administration; Bioven; Coronavirus
MeSH Terms: conditions — COVID-19; Pneumonia; Coronavirus Infections | interventions — Immunoglobulins, Intravenous; gamma-Globulins; Administration, Intravenous

STUDY DESIGN:
Intervention Model Description: Open-label multicenter randomized controlled in parallel groups.
  Patients undergoing screening are randomized into groups in equal proportions:
  * Study Group (receive IVIG Bioven with base therapy).
  * Control group (receive base therapy only)
  At the stage of Data Analysis to ensure comparability of data and homogeneity of the sample, the possibility of additional comparison of groups based on the actually prescribed base therapy and other identified covariates is provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (IVIG) (Experimental): Patients receive IVIG (trade name - Bioven) with base therapy
  Interventions: Drug: IVIG
- Control group (No Intervention): Patients receive base therapy only

INTERVENTIONS:
Drug: IVIG — Patients in the study group receive the drug Bioven, 10% solution for infusions produced by LLC Biopharma Plasma 0,8-1,0 g/kg once a day for 2 days (total course dose - 1.6-2.0 g/kg) as well as base treatment recommended by the protocol of COVID-19 coronavirus infection treatment depending on the severity of their condition according to the prescription sheet.
  Other Names: Human normal immunoglobulin for intravenous administration; Bioven
  Arms: Study Group (IVIG)

SUMMARY:
Pneumonia caused by coronavirus infection COVID-19 is characterized by a combination of several dangerous factors that consistently worsen the patient's condition: viral lung damage early in the disease; a sharp increase in inflammation on the background of an unbalanced immune response ("cytokine storm"); joining a bacterial infection.

The condition of patients deteriorates significantly mostly at cytokine storm development. The damaging of a large volume of lung tissue leads to develops of respiratory failure, respiratory distress syndrome, or shock. Ventilatory support becomes ineffective and patients die.

There are reports of the effectiveness of Human Normal Immunoglobulin for Intravenous Administration (IVIG) high doses when used as part of complex therapy in patients with pneumonia caused by coronavirus COVID-19. In particular, IVIG has a positive effect on survival rates, overall disease course, duration of stay in the intensive care unit, and ventilatory support duration.

The probable mechanism of action of high-dose IVIG therapy is considered to be a regulatory effect on the immune system. Similar is the known and confirmed effectiveness of IVIG for autoimmune diseases (Kavasaky disease, Guillain Barre syndrome, Chronic inflammatory demyelinating polyradiculoneuropathy, Multifocal motor neuropathy).

This trial to assesses the Efficacy of IVIG (medication trade name - Bioven, manufactured by Biopharma Plasma LLC) in the High Immunomodulatory Dose in Complex Treatment of Severe Pneumonia Caused by COVID-19 / SARS-CoV-2

DETAILED DESCRIPTION:
The screening stage:

The patient or his legal representative must sign an informed consent. After signing the informed consent, the screening tests&procedures are performed and the compliance with the inclusion / non-inclusion criteria is assessed.

For patients who have been screened and meet the inclusion criteria and do not fall under the exclusion criteria, a blinded randomization procedure is provided.

Randomization is performed by the IVRS method, according to the blinded-block patient's randomization table.

The clinical stage of the trial:

Begins after patient randomization. At the clinical stage, among other things, provides:

* Determination of the individual dose of the study drug (in the study group)
* Administration of the drug (in the study group)
* Registration of adverse events
* registration of information about taking antiviral drugs for the treatment of COVID-19;
* registration of information on symptomatic therapy and administration of drugs for the treatment of comorbidities;
* measurement of vital signs (blood pressure, heart rate, respiratory rate, body temperature);
* Determination of SPO2 level
* Determining the need for ventilation
* Determining the need for intensive care
* Assessment of compliance with the exclusion criteria

Patients in the Control Group will receive therapy recommended by the COVID-19 coronavirus infection treatment protocol, depending on the severity of their condition according to the prescribing list, which will not include immunoglobulin preparations.

Patients of the Study Group (IVIG) receive high-dose therapy with the study drug (Bioven, 10% solution for infusions produced by Biopharma Plasma LLC, Ukraine). The dose is calculated by body weight. Patients will also receive therapy recommended by the COVID-19 coronavirus infection treatment protocol, depending on the severity of their condition according to the prescribing list.

Bioven administered intravenously, at an initial rate of 0.5 - 1.0 ml/kg body weight/hour for 30 minutes. In the absence of any undesirable side effects, the rate of administration can be gradually increased (recommended increase by 0.5 - 1.5 ml/kg body weight/hour every 10 minutes). According to results previously accomplished clinical studies, the maximum rate of Bioven administration is up to 8.5 ml/kg body weight/hour.

Observation and completion stage:

Begins and continues from the last administration of the study drug until the discharge of the patient from the hospital, but not less than 28 days from the confirmation of the diagnosis of pneumonia caused by coronavirus infection COVID-19.

The following procedures are provided at the stage:

* registration of information about taking antiviral drugs for the treatment of COVID-19;
* registration of information on symptomatic therapy and administration of drugs for the treatment of comorbidities;
* measurement of vital signs (blood pressure, heart rate, respiratory rate, body temperature);
* determination of SPO2 level
* registration of the results of the examination of the lungs by computed tomography (or radiography)
* taking biomaterials for laboratory research:
* general blood test (erythrocytes, hemoglobin, expanded leukocyte formula, platelets, etc.);
* general analysis of urine;
* biochemical analysis of blood;
* state of the coagulation system
* determination of inflammatory factors in the dynamics (CRP, ferritin, procalcitonin; TNF-α), IL-1-beta, IL-6, complement component C3 (C3), circulating immune complexes (CIC), etc.),
* determination of IgG subclasses (G1, G2, G3, G4,);
* Determining the need for ventilation
* Determining the need for intensive care
* Adverse reactions registration
* Assessment of compliance with the exclusion criteria

The patient's condition is assessed daily till discharge; and by schedule after discharge (if it happen earlier), during 28 days period after diagnosis of severe pneumonia caused by coronavirus infection COVID-19 In case of death of the patient - the date and cause of death are fixed. The results of the study are evaluated by endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years of age and older;
* COVID-19 documentary confirmed by PCR lab test;
* severe pneumonia caused by COVID-19 according to the criteria below:

  * - fever or suspicion of respiratory infection;
  * - the number of respiratory movements 30 per 1 min and above;
  * - severe respiratory failure or SpO2 <90% with spontaneous breathing indoors;
  * - the presence of foci of inflammation in the lungs according to the results of computed tomography, which is documented.
  * or if any of the conditions listed below have developed on the background of previously diagnosed coronavirus pneumonia:

    * - severe respiratory failure required mechanical ventilation (ALV);
    * - acute respiratory distress syndrome according to WHO diagnostic criteria (development within one week after the manifestation of disease clinical symptoms or emergence of new ones or deterioration of respiratory syndromes. Chest visualization (lung X-ray, CT or ultrasound); bilateral opacities not fully explaining the gravity of condition or lung collapse or nodules);
    * - sepsis according to WHO diagnostic criteria (life-threatening organ dysfunction caused by disturbance of host reaction to suspected or proven infection. The features of organ dysfunction include the following: mental change, labored or shallow breathing, low oxygenation, oliguria or anuria, rapid heart palpitation, weak pulse, cold extremities or low blood pressure, skin blotching or lab-proven coagulopathy, thrombocytopenia, acidosis, high level of lactic acid or hyperbilirubinemia);
    * - endotoxic shock according to WHO diagnostic criteria (persisting hypotension despite extensive resuscitation requiring vasoconstrictors for maintaining mean arterial pressure ≥ 65 mmHg and serum lactate level > 2 mmol/l);
* the signed patient's informed consent to participation in the trial;
* the negative pregnancy test (for female patients of reproductive age), readiness to use reliable contraception methods during the whole duration of the trial.
* the ability, according to the researcher, to follow all requirements of the research protocol.
* this study allows you to take into account the results of examinations related to the disease, conducted within 10 days before signing the Informed Consent. Such data are transferred from the primary documentation to the CRF.

Exclusion Criteria:

* known intolerance to plasma or immunoglobulin drugs;
* drug allergy or hypersensitization to immunoglobulin drugs;
* any known counter-indication to immunoglobulin drugs according to the instruction for medical application of the tested drug;
* pneumonia not associated with COVID-19 infection;
* pregnancy, lactation period;
* any clinically significant impairment of liver function (elevation of serum transaminase levels more than 3 times the upper limit of normal);
* serum creatinine levels more than 2 times the upper limit of normal for a given age and gender;
* established diagnosis of primary immunodeficiency;
* verified HIV-infection;
* immune diseases (blood immune diseases, rheumatic diseases, nephritis, etc.)
* severe cardiovascular failure (Stage III);
* mental illness in anamnesis;
* the need for prescribing medicines or procedures that are incompatible with the administration of the drug within the scope of this study: monoclonal antybodies;
* known drug addiction;
* participation in any other clinical trial presently or within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Period duration (in days) to clinical improvement | From date post-onset of severe pneumonia to date of patient discharge or date of death, whichever came first, assessed up to 28 days
  Number of days post-onset of severe pneumonia to the moment of normalization at least two from following primary outcomes: O2 saturation with self-breathing, respiratory movements rate with self-breathing, body temperature without antipyretics use, lymphocyte count (targeted levels set in the description each of these primary outcomes)
O2 saturation (SPO2 percentage), with self-breathing | From date post-onset of severe pneumonia to date of patient discharge or date of death, whichever came first, assessed up to 28 days
  The target level of SPO2 percentage - 95% and above with self-breathing, is used as one of the clinical improvement criteria
Respiratory movements rate (amount per minute), with self-breathing | From date post-onset of severe pneumonia to date of patient discharge or date of death, whichever came first, assessed up to 28 days
  The target level of respiratory movements - 28 per minute or less with self-breathing, is used as one of the clinical improvement criteria
Body temperature without antipyretics use | From date post-onset of severe pneumonia to date of patient discharge or date of death, whichever came first, assessed up to 28 days
  Measured in degrees Celsius. Fever absence (body temperature no more 37 degrees Celsius) during at least 24 hours without antipyretics, is used as one of the clinical improvement criteria.
Lymphocyte count | From date post-onset of severe pneumonia to date of patient discharge or date of death, whichever came first, assessed up to 28 days
  The target level 1000 cells / mm3 and above is used as one of the clinical improvement criteria (applicable for patients with lymphocytes count lower 1000 cells / mm3 at screening moment)

SECONDARY OUTCOMES:
Time from the onset of the disease to discharge, in days | 28 days
  Period duration (in days)
Duration of the need for ventilatory support, in days | 28 days
  Number of days with ventilatory support
Duration of the need for intensive care, in days | 28 days
  Number of days in the intensive care unit
Duration of need for oxygenation in days (SPO2 ≤ 93% with self-breathing) | 28 days
  Number of days with necessery of oxygenation support
The C-reactive protein (CRP) level | Day 0 (screening), day 5, day 14, day 28
  Measuring the analyte concentration in plasma (mg/L)
The tumor necrozis factor alpha (TNF-α) level | Day 0 (screening), day 5, day 14, day 28
  Measuring the analyte concentration in plasma (pg/mL)
The interleukin-1β (IL-1β) level | Day 0 (screening), day 5, day 14, day 28
  Measuring the analyte concentration in plasma (pg/mL)
The interleukin-6 (IL-6) level | Day 0 (screening), day 5, day 14, day 28
  Measuring the analyte concentration in plasma (pg/mL)
The D-dimer level | Day 0 (screening), day 5, day 14, day 28
  Measuring the analyte concentration in plasma (µg FEU/mL)
The Complement (C3 component) level | Day 0 (screening), day 5, day 14, day 28
  Measuring the analyte concentration in plasma (g/L)
The Circulating immune complexes level | Day 0 (screening), day 5, day 14, day 28
  Measuring the analyte concentration in plasma (U/mL)
The ferritin level | Day 0 (screening), day 5, day 14, day 28
  Analyte concentration in plasma (ng/mL)
The procalcitonin level | Day 0 (screening), day 5, day 14, day 28
  Analyte concentration in plasma (ng/mL)
IgG subtypes | Day 0 (screening), day 5, day 14, day 28
  The IgG-subtypes (IgG1-IgG4) concentration in plasma (mg/dL)
Survival assessment for a 28-day follow-up period since the onset of severe pneumonia | 28 days
  Survivealance estimation

OTHER OUTCOMES:
Frequency of side effects | 28 days
  Number of participants with adverse reactions related by investigational drug as assessed by CTCАЕ v 4.0
Frequency of serious side effects | 28 days
  Number of participants with serious adverse reactions related by investigational drug as assessed by CTCАЕ v 4.0

CONTACTS AND LOCATIONS:
Locations (9):
- Ukraine (9):
  - Site 08 - "Central City Clinical Hospital of Ivano-Frankivsk City Council", Ivano-Frankivsk, Ivano-Frankivs'k Region
  - Site 02 - "Bila Tserkva City Hospital №3", Bila Tserkva, Kyiv Oblast
  - Site 03 - "Lviv Regional Infectious Diseases Clinical Hospital", Lviv, Lviv Oblast
  - Site 04 - "City Clinical Infectious Diseases Hospital", Odesa, Odesa, Odesa Oblast
  - Site 07 - "Ternopil City Municipal Ambulance Hospital", Ternopil, Ternopil Oblast
  - Site 06 - "Vinnytsia City Clinical Hospital №1", Vinnitsia, Vinnitsia Region
  - Site 09 - "Volyn Regional Clinical Hospital", Lutsk, Volyn Oblast
  - Site 01 - "Kyiv City Clinical Hospital №17", Kyiv
  - Site 05 - "Kyiv City Clinical Hospital №4", Kyiv

IPD SHARING:
Plan to Share IPD: Yes
After completion of the trial, results will be published. Access to parts CSR planned after the release of scientific publications
Supporting Information: CSR
Time Frame: After trial result publication 3 months later
Access Criteria: For specialists in medicine, pharmacy, scientists